CLINICAL TRIAL: NCT01960608
Title: The Analysis of Correlation About the Spot Urine Sodium and the Blood Pressure in General Population According to the Income Level
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Hoseok Koo, Assisted professior, Inje University
Other Study IDs: sodium_income
Record Dates: First submitted 2013-10-06; First posted 2013-10-10 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (7):
- low sodium group: 24_hours_urine_sodium < 100 mEq/L
  Interventions: Other: 24_hours_urine_sodium
- mid sodium group: 24_hours_urine_sodium >= 100 mEq/L and < 200 mEq/L
  Interventions: Other: 24_hours_urine_sodium
- high sodium group: 24_hours_urine_sodium >= 200 mEq/L
  Interventions: Other: 24_hours_urine_sodium
- low income group: the income 25% below the quartile
- low mid income group: the income 25% - 50% below the quartile
- mid income group: the income 50% - 75% below the quartile
- high income group: the income 75% over the quartile

INTERVENTIONS:
Other: 24_hours_urine_sodium
  Groups: high sodium group; low sodium group; mid sodium group

SUMMARY:
Increasing sodium intake raises blood pressure. And high salt intake could hinder the management of chronic disease. Much previous research has confirmed that dietary habits are affected by economic status. So we compared sodium intake with economic status. We investigated the prevalence, extent and management, and the relevance of sodium intake with income level.

ELIGIBILITY:
Inclusion Criteria:

* all the patient who participated in the national survey

Exclusion Criteria:

* no pregnancy
* malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general population
Sampling Method: Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
sodium intake and the degree of control of blood pressure in general population according to the income level | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Seoul Paik Hospital, Seoul, Seoul, South Korea